CLINICAL TRIAL: NCT01102608
Title: Phase II Study of Neoadyuvant High-dose Ifosfamide and Concurrent Radiotherapy in Soft Tissue Sarcoma and Identification of Response Predictors
Brief Title: Neoadyuvant High-dose of Ifosfamide and Concurrent Radiotherapy in Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Principal Investigator, Mariló de Carrillo, Dr. Xavier García del Muro, Grupo Espanol de Investigacion en Sarcomas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS15; Nº EudraCT:2007-005755-42
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: sarcoma; ifosfamide
MeSH Terms: conditions — Sarcoma | interventions — Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Ifosfamide

INTERVENTIONS:
Drug: Ifosfamide — 3 cycles of Ifosfamide (12g/m2) associated to Mesna (6g/m2), in i.v infusion 6 days, every 3 weeks

SUMMARY:
To study the activity and toxicity of a neoadjuvant regimen including high-dose ifosfamide in combination with radiotherapy, and subsequent surgery, in high-risk soft tissue sarcomas.

DETAILED DESCRIPTION:
This is a phase II multicenter study designed in two phases. A total of 32 patients will be included in 10 hospitals belonging to the Spanish Group for Research in Sarcomas (GEIS). Selection criteria are: patients with localized soft tissue sarcoma from the extremities or trunk with high-risk features (>5 cm and grade 2-3), or recurrences after prior inadequate surgery. The treatment schedule will be: initial biopsy, 3 cycles of high-dose Ifosfamide, 12 gr/m2 in 5 days, concurrent with Radiotherapy 50 Gy, and subsequent wide surgery. To assess the predictive factors of response to the combination therapy, DNA and RNA extraction will be performed on the pretreatment biopsies. DNA will be used to hybridize Affymetrix GeneChip® Human Mapping 500K Array, which allows for the study of 500000 SNPs throughout the genome. The expression of 39000 RNA transcripts will be evaluated employing the Affymetrix Genechip Human Genome HG-U133 Plus 2.0, and validated by real-time RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Advanced Soft Tissue Sarcoma histological proven, potentially resected, located in extremities and trunk for one of the following histological subtypes: leiomyosarcoma, undifferentiated pleomorphic sarcoma, Synovial Sarcoma, Liposarcoma and malignant tumour of peripheral nerve sheath.
2. Primary tumour:

   1. Size ³ 5 cm of diameter
   2. Histological grade 2-3
   3. Deep location
3. No distant metastases
4. Patients must have not been previously treated with Chemotherapy or Radiotherapy on the tumour area.
5. However patients are eligible with local relapse after previous surgery.
6. Patients must be £18 and ³ 65 years old.
7. Patients must have ECOG performance status 0 to 1
8. Patients must have measurable disease by Recist Criteria.
9. Absolute neutrophil count ³1,500/mm3, platelet count ³ 100,060 ml/min, creatinine, total bilirubin, ALT and AST £ 1.5 times the upper limit of normal
10. Signed informed consent prior to any study specific procedures

Exclusion Criteria:

1. Patients with cerebral metastasis
2. Pregnant or breast feeding patients.
3. Active infection or other concomitant severe illness.
4. Severe psychiatric illness which would not make possible the obtention of the informed consent
5. Concurrent treatment with other experimental drugs within 30 days prior to study entry.
6. History of previous treated or diagnosed cancer in the past 5 years, excepting basocellular cell skin cancer, cervix cancer in situ or superficial bladder carcinoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of the neoadyuvant high-dose of ifosfamide and radiotherapy, determined with clinical and pathological responses | 10 weeks since the inclusion of the patient

SECONDARY OUTCOMES:
Global survival, free relapse survival and toxicity | Until relapse or patient´s death

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro, Doctor, Study Chair — Grupo Español de Investigacion en Sarcomas
Locations (1):
- Grupo Espanol de Investigación en Sarcomas, Barcelona, España, Spain

REFERENCES:
- See also: Related Info — http://www.grupogeis.org